CLINICAL TRIAL: NCT01077934
Title: Assessment of Near Infrared Spectroscopy as a Diagnostic Tool in Acute Compartment Syndrome
Status: Completed | Type: Observational
Sponsor: J&M Shuler (Industry)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, William Reisman, Principal Investigator, Emory University
Other Study IDs: 01-10-14b
Record Dates: First submitted 2010-02-24; First posted 2010-03-01 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Compartment Syndrome
Keywords: All Patients admitted to Grady Memorial Hospital with Unilateral Lower leg injury at risk for compartment syndrome
MeSH Terms: conditions — Compartment Syndromes | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Injured Extremity without compartment syndrome
  Interventions: Device: near-infrared spectroscopy
- Injured extremity with compartment syndrome
  Interventions: Device: near-infrared spectroscopy

INTERVENTIONS:
Device: near-infrared spectroscopy — Non-invasive monitoring device applied on the surface of the skin that emits harmless red light to measure tissue perfusion.

SUMMARY:
The purpose of this study is to define the reliability and accuracy of Near Infrared Spectroscopy (NIRS) in the detection of intra-compartmental tissue perfusion in injured and noninjured extremities over time. We hypothesize that this technology, combined with vital signs, intracompartmental pressures and clinical examinations, will be useful in diagnosing acute compartment syndrome (ACS), monitoring patients at risk for ACS, and evaluating the adequacy of fasciotomy in patients treated for ACS.

DETAILED DESCRIPTION:
Acute compartment syndrome (ACS) is associated with lower leg trauma in up to 20% of high energy injuries. ACS occurs when the pressure due to swelling exceeds the perfusion pressure thereby cutting off blood flow to the leg. If untreated, the results can be catastrophic with an insensate, contracted leg. Moreover, there is a high risk of subsequent infection and even amputation. The treatment for ACS, a four compartment fasciotomy, is aimed at releasing the pressure through two incisions from roughly the knee to the ankle. Often due to wound expansion, the incisions require multiple debridements and skin grafting to close. With fasciotomies, fractures are converted from closed to open injuries. When left open for many days, the risk of infection and complications such as nonunion increase significantly.

The only accepted objective method for diagnosis of ACS is to measure the pressure inside the leg compartments by using a large gauge needle hooked to a pressure monitor. However, these readings can be erroneous if not performed correctly. As such, ACS continues to be a clinical diagnosis which is made based on the surgeon's experience and their interpretation of the character of the injury (high-energy, motorcycle crash, vs. low-energy, a twisted ankle). Clinicians are left to attempt to interpret physical exam findings and readings from pressure monitors. Most importantly ACS is not an event, but a process that can manifest at multiple points after injury. The most accurate and effective method for diagnosing and appropriately treating ACS is serial examination over a course of hours to days.

With this study, we hope to evaluate the NIRS device, which is non-invasive, as diagnostic tool in the evaluation of acute compartment syndrome. We plan to evaluate all patients by the gold standard in diagnosing acute compartment syndrome while simultaneously evaluating the patient with the NIRS device. This will allow us to determine if the NIRS device can accurately and reliably predict the development of acute compartment syndrome in a non-invasive, longitudinal manner.

"Access to a precise, reliable, and noninvasive method for early diagnosis of ACS would be a landmark achievement in orthopaedic and emergency medicine."

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included between the ages of thirteen and eighty-five who are willing to participate and have unilateral lower leg injury with a fracture to the tibia.

Exclusion Criteria:

* Patients will be excluded from enrollment if they have bilateral injuries to the lower legs or have been previously diagnosed peripheral vascular disease. Patients will also be excluded if they are not willing to participate.

Ages: 13 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Patients admitted to Grady with Unilateral Lower leg injury at risk for compartment syndrome
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
NIRS values in lower leg extremity injury | 4 days
  We will monitor patients during their hospital stay from the time of admission until discharge at likey day 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States